CLINICAL TRIAL: NCT06170333
Title: Efficacy and Side Effects of 8% Sulphur-Aloe Vera Soap Versus Bland Soap as an Adjuvant of Ketoconazole 2% Shampoo for the Treatment of Pityriasis Versicolor: Open Controlled Trial
Brief Title: 8% Sulphur-Aloe Vera Soap as an Adjuvant Treatment for Pityriasis Versicolor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV-202309.02
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pityriasis Versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — Sulfur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8% sulphur and A. vera soap and ketoconazole 2% shampoo (Experimental): Twenty-one patients will be given the combination of 8% sulphur and A. vera soap applied to the entire body surface (excluding face), left on for five minutes and then washed off. This was applied twice daily for four weeks.
  Along with the soap or placebo, patients will receive 2% ketoconazole shampoo, left on for five minutes and then washed off. This was applied thrice weekly for a week
  Interventions: Drug: 8% sulphur and A. vera soap
- Bland soap and ketoconazole 2% shampoo (Active Comparator): Twenty-one patients will be given bland soap applied to the entire body surface (excluding face), left on for five minutes and then washed off. This was applied twice daily for four weeks.
  Along with the soap or placebo, patients will receive 2% ketoconazole shampoo, left on for five minutes and then washed off. This was applied thrice weekly for a week.
  Interventions: Drug: 8% sulphur and A. vera soap

INTERVENTIONS:
Drug: 8% sulphur and A. vera soap — Patients in experimental arms will receive the combination of 8% sulphur and A. vera soap for four weeks along with 2% ketoconazole shampoo for a week.
  Other Names: Blacksoap

SUMMARY:
Pityriasis versicolor (PV) is a superficial, mild, often chronic recurring infection of the skin caused by Malassezia species which is characterized by the formation of hypopigmented, hyperpigmented and/or erythematous macules. It commonly occurs on the trunk and proximal extremities, but can also be found on the entire body. Diagnosis of PV established based on clinical features and microscopic examination with potassium hydroxide. The goals of PV treatment are: to eradicate the hyphae, disappearance of clinical signs and symptoms, to lessen recurrences, and improve patient's quality of life. Topical antifungal remains first line therapy and search for an ideal topical agent of PV continue. Various studies reported combining more than one topical agents can increase the efficacy, thus result in faster mycological cure.

DETAILED DESCRIPTION:
Pityriasis versicolor commonly has extensive and irregular pattern/distribution on the body. Therefore, topical antifungal such as ketoconazole, usually given in shampoo or solution form to cover large surface area. Many studies reported adverse effects of ketoconazole shampoo including pruritus, dry skin, and allergic contact dermatitis. Non-spesific keratolytic agent, such as sulphur, used for PV work by desquamation of the entire superficial skin layer and eliminating the fungi in the process. It also could enhance the penetration of ketoconazole into the stratum corneum, increasing its potency. Aloe vera (A. vera) contains acetylated mannan that acts as humectant and increase water content in stratum corneum. The combination of sulphur and A. vera in form of a soap as adjuvant to ketoconazole shampoo potentially will result in synergistic effect, faster mycological cure, and less adverse effects. There are limited data of sulphur and A.vera soap as an adjuvant PV treatment to ketoconazole shampoo. As a result of limited data, our trial is looked forward to assess the efficacy and adverse effect of sulphur and A.vera soap as an adjuvant PV treatment to ketoconazole shampoo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-65 years
3. Diagnosed as PV based on clinical features, microscopic examination using 10% potassium hydroxide, and Wood's lamp

Exclusion Criteria:

1. Pregnant or lactating women
2. PV with concurrent skin conditions (dermatitis or skin lesions in form of vesicles or blister or pustules or erosions or excoriation) with body surface area >30%
3. Use of topical antifungal and/or corticosteroid 14 days prior to study entry
4. Use of systemic antifungal and/or corticosteroid 30 days prior to study entry
5. History of allergy to shampoo or soap containing ketoconazole, sodium lauryl sulphate, sulphur, A. vera, charcoal powder, glycerin, or perfume.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of pruritus | 28 days
  A visual analogue score (VAS) will be used to assess pruritus according to the following scale: 0 = no pruritus; 1-3 = mild pruritus; 4-6 = moderate pruritus; 7-10 = severe pruritus.
Scaling severity | 28 days
  Patients will be evaluated for scaling severity according to the following scale: 0 = no scaling; 1 = mild distribution of scaling; 2 = moderate distribution of scaling; 3 = severe, extensive distribution of scaling.
Mycological cure | 28 days
  Evaluation of mycological cure examined by microscopic examination using 10% potassium hydroxide. A cellophane tape will be used for taking scale lesions.

SECONDARY OUTCOMES:
Wood's lamp | 28 days
  Fluorescence of skin lesions using Wood's lamp will be evaluated every visit. Positive result obtained if skin lesions showed yellow fluorescence.
Skin hydration | 28 days
  Skin hydration will be measured using corneometer on three areas: volar, wrist, and palms. Scores are expressed in arbitary units (AU), AU <30 means very dry skin, AU between 30 -40 means dry skin, and AU >40 means normal skin
Skin pH (potential hydrogen) | 28 days
  Skin pH will be measured using pH on three areas: volar, wrist, and palms. Normal skin pH values range from pH 4.0 to 7.0. pH level below 7 considered acidic and above 7 considered alkaline.

CONTACTS AND LOCATIONS:
Overall Officials: Risa Miliawati Nurul Hidayah, MD, Ph.D, Principal Investigator — Faculty of Medicine, Universitas Padjadjaran, Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia